CLINICAL TRIAL: NCT00087607
Title: A Prospective, Randomized, Open-label Study Evaluating the Viral Kinetics and Pharmacokinetics of Pegasys® Plus Copegus® and PEG-Intron® Plus Rebetol® in Interferon-naïve Patients With Chronic Hepatitis C.
Brief Title: Peak Study - A Study of Pegasys (Peginterferon Alfa-2a (40KD)) in Combination With Copegus (Ribavirin) in Interferon-Naive Patients With Chronic Hepatitis C (CHC).
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML17756
Record Dates: First submitted 2004-07-12; First posted 2004-07-14 (Estimated); Results first posted 2016-07-01 (Estimated); Last update posted 2016-07-01 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — Ribavirin; peginterferon alfa-2b; peginterferon alfa-2a

ARMS (2):
- Peginterferon Alfa-2a + Ribavirin (Experimental): Participants received Peginterferon alfa-2a (40 kD) [Pegasys] at a dosage of 180 microgram (μg), subcutaneously (SC), once a week plus Ribavirin [Copegus] 1000 or 1200 milligram (mg)/day), orally, [according to body weight, lesser than or greater than/equal to (< or >/=) 75 kilogram (kg), respectively] twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a 180 μg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
  Interventions: Drug: Ribavirin; Drug: Peginterferon alfa-2a [Pegasys]
- Peginterferon Alfa-2b + Ribavirin (Active Comparator): Participants received Peginterferon alfa-2b (12 kD) [PEG-Intron] at a dosage of 1.5 μg/kg SC once weekly plus Ribavirin [Rebetol] 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a 180 μg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
  Interventions: Drug: Peginterferon alfa-2b (PEG-Intron); Drug: Ribavirin

INTERVENTIONS:
Drug: Ribavirin — 1000/1200mg/day po
  Other Names: Copegus
  Arms: Peginterferon Alfa-2a + Ribavirin
Drug: Peginterferon alfa-2b (PEG-Intron) — 1.5 micrograms/kg sc weekly
  Arms: Peginterferon Alfa-2b + Ribavirin
Drug: Ribavirin — 1000/1200mg/day po
  Other Names: Rebetol
  Arms: Peginterferon Alfa-2b + Ribavirin
Drug: Peginterferon alfa-2a [Pegasys] — 180 micrograms sc weekly
  Arms: Peginterferon Alfa-2a + Ribavirin

SUMMARY:
This study will examine the viral kinetics and pharmacokinetics of Pegasys plus ribavirin and PEG-Intron plus ribavirin in interferon-naive patients with CHC. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients at least 18 years of age
* CHC infection, genotype 1
* use of 2 forms of contraception during study in both men and women

Exclusion Criteria:

* previous systemic therapy with anti-viral, anti-neoplastic, or immunomodulatory agents
* medical condition associated with chronic liver disease (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposure)
* decompensated liver disease
* women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2004-01; Primary Completion 2006-03 (Actual); Study Completion 2006-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (39):
- United States (39):
  - Birmingham, Alabama
  - Little Rock, Arkansas
  - Sacramento, California
  - San Diego, California
  - San Francisco, California
  - San Mateo, California
  - San Rafael, California
  - Farmington, Connecticut
  - Hartford, Connecticut
  - Bradenton, Florida
  - Miami, Florida
  - Wellington, Florida
  - Kansas City, Kansas
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - Detroit, Michigan
  - Kansas City, Missouri
  - St Louis, Missouri
  - Omaha, Nebraska
  - Las Vegas, Nevada
  - East Orange, New Jersey
  - Egg Harbour Township, New Jersey
  - Vineland, New Jersey
  - New York, New York
  - Poughkeepsie, New York
  - The Bronx, New York
  - Fayetteville, North Carolina
  - Statesville, North Carolina
  - Portland, Oregon
  - Columbia, South Carolina
  - Austin, Texas
  - Dallas, Texas
  - Fairfax, Virginia
  - Norfolk, Virginia
  - Roanoke, Virginia
  - Tacoma, Washington
  - Racine, Wisconsin

REFERENCES:
- [Derived] Chung RT, Poordad FF, Hassanein T, Zhou X, Lentz E, Prabhakar A, Di Bisceglie AM. Association of host pharmacodynamic effects with virologic response to pegylated interferon alfa-2a/ribavirin in chronic hepatitis C. Hepatology. 2010 Dec;52(6):1906-14. doi: 10.1002/hep.23947. Epub 2010 Nov 9. PMID 21064034
- [Derived] Di Bisceglie AM, Ghalib RH, Hamzeh FM, Rustgi VK. Early virologic response after peginterferon alpha-2a plus ribavirin or peginterferon alpha-2b plus ribavirin treatment in patients with chronic hepatitis C. J Viral Hepat. 2007 Oct;14(10):721-9. doi: 10.1111/j.1365-2893.2007.00862.x. PMID 17875007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from January 2004 to April 2006 at 41 centers in the United States.
Pre-assignment Details: This study planned to enroll 344 participants (172 in each group). Of the total randomized 385 participants who met the eligibility criteria, five did not receive study treatment and were not included in any analysis population.
Period: Overall Study
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Started | 192 | 193
Completed | 70 | 71
Not Completed | 122 | 122
Not completed — Adverse Event | 14 | 24
Not completed — Death | 0 | 1
Not completed — Insufficient Therapeutic Response | 53 | 42
Not completed — Failure to return | 21 | 17
Not completed — Withdrew Consent | 12 | 16
Not completed — Administrative | 12 | 12
Not completed — Refused Treatment | 5 | 7
Not completed — Other Protocol Violation | 5 | 2
Not completed — Violation of Selection Criteria at Entry | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were described for the Intent-to-Treat (ITT) Population, which included all participants who were randomized and received at least one dose of study medication (Pegylated interferon [PEG-IFN] or ribavirin).
Groups:
- Peginterferon Alfa-2a + Ribavirin: Participants received Peginterferon alfa-2a at a dosage of 180 μg SC once a week plus Ribavirin 1000 or 1200 mg/day, orally (< or >/= 75 kg body weight, respectively) twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a 180 μg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
- Peginterferon Alfa-2b + Ribavirin: Participants received Peginterferon alfa-2b at a dosage of 1.5 μg/kg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a 180 μg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin | Total
Number analyzed (Participants) | 189 | 191 | 380
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.9 (7.18) | 48.4 (7.80) | 47.6 (7.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 55 | 123
  Male | 121 | 136 | 257

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Viral Load (log10 Reduction) at Week 12
Description: The viral load was determined quantitatively and qualitatively by Hepatitis C virus (HCV)-polymerase chain reaction (PCR). HCV RNA was measured qualitatively using the Roche amplicor PCR assay (lower limit of detection 60 international units per milliliter (U/mL), changed from 50 IU/mL with amendment B) and quantitatively using the Roche amplicor HCV monitor® test v2.0 (lower limit of quantification 600 IU/mL). Log transformations were performed for HCV RNA, and the analyses were done on a log10 scale. The average value of the difference between viral load levels in the serum from baseline to Week 12, expressed in terms of a logarithmic scale with base 10, are presented.
Time Frame: From Baseline to Week 12
Population: The analysis population was ITT Population. The ITT Population included all participants who were randomized and received at least one dose of study medication (PEG-IFN or ribavirin). Data using ITT Population are presented below.
Measure: Mean (Standard Error); unit: log (IU/mL)
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 172 | 169
log (IU/mL) | -3.26 (0.12) | -3.27 (0.14)
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Mean treatment difference was tested using a two-sided t-test; Test type: Superiority or Other; p = 0.978, t-test, 2 sided; Mean Difference (Net) = 0.01, 95% CI 2-sided [-0.35 to 0.36]

2. Secondary Outcome: Mean Change From Baseline in Viral Load (log10 Reduction) at Week 4 and Week 8
Description: The viral load was determined quantitatively and qualitatively by HCV-PCR. HCV RNA was measured qualitatively using the Roche amplicor PCR assay (lower limit of detection 60 IU/mL, changed from 50 IU/mL with amendment B) and quantitatively using the Roche amplicor HCV monitor® test v2.0 (lower limit of quantification 600 IU/mL). Log transformations were performed for HCV RNA, and the analyses were done on a log10 scale. The average value of the difference between viral load levels in the serum from baseline to week 4 and week 8, expressed in terms of a logarithmic scale with base 10 are presented.
Time Frame: Baseline, Week 4 and Week 8
Population: The analysis population was ITT Population. The ITT Population included all participants who were randomized and received at least one dose of study medication (PEG-IFN or ribavirin).The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Error); unit: log (IU/mL)
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 181 | 178
log (IU/mL)
  Week 4; n = 181, 178 | -1.95 (0.10) | -2.22 (0.12)
  Week 8; n = 178, 175 | -2.88 (0.12) | -2.95 (0.13)
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; At Week 4: Mean treatment difference was tested using a two-sided t-test; Test type: Superiority or Other; p = 0.080, t-test, 2 sided; Mean Difference (Net) = 0.27, 95% CI 2-sided [-0.03 to 0.58]
Statistical Analysis 2: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; At Week 8: Mean treatment difference was tested using a two-sided t-test; Test type: Superiority or Other; p = 0.688, t-test, 2 sided; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.27 to 0.41]

3. Secondary Outcome: Weekly Viral Load Assessed at Drug Trough
Description: The viral load was determined quantitatively and qualitatively by HCV-PCR. HCV RNA was measured qualitatively using the Roche amplicor PCR assay (lower limit of detection 60 IU/mL, changed from 50 IU/mL with amendment B) and quantitatively using the Roche amplicor HCV monitor® test v2.0 (lower limit of quantification 600 IU/mL). Log transformations were performed for HCV RNA, and the analyses were done on a log10 scale. The viral load levels in the serum at baseline and for each week, were expressed in terms of a logarithmic scale with base 10, and averaged for all participants.
Time Frame: Baseline, up to Week 12
Population: The analysis population was ITT Population. The ITT Population included all participants who were randomized and received at least one dose of study medication (PEG-IFN or ribavirin). The "n" represents the number of participants analyzed at a specified time point.
Measure: Mean (Standard Deviation); unit: log (IU/mL)
Groups:
- Peginterferon Alfa-2a + Ribavirin: Participants received Peginterferon alfa-2a at a dosage of 180 μg SC once a week plus Ribavirin 1000 or 1200 mg/day, orally (< or >/= 75 kg body weight, respectively) twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a180 μg SC once weekly plus Ribavirin1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
- Peginterferon Alfa-2b + Ribavirin: Participants received Peginterferon alfa-2b at a dosage of 1.5 μg/kg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a180 μg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 189 | 191
log (IU/mL)
  Baseline; n = 189, 191 | 6.46 (0.35) | 6.48 (0.37)
  Week 1; n = 181, 185 | 5.69 (0.87) | 5.70 (0.89)
  Week 2; n = 182, 184 | 5.26 (1.11) | 5.12 (1.25)
  Week 3; n = 179, 183 | 4.84 (1.31) | 4.64 (1.47)
  Week 4; n = 181, 178 | 4.51 (1.42) | 4.25 (1.57)
  Week 5; n = 182, 179 | 4.20 (1.48) | 4.01 (1.61)
  Week 6; n = 179, 177 | 3.96 (1.53) | 3.78 (1.66)
  Week 7; n = 178, 175 | 3.73 (1.54) | 3.64 (1.67)
  Week 8; n = 178, 175 | 3.57 (1.55) | 3.53 (1.67)
  Week 9; n = 171, 170 | 3.44 (1.56) | 3.44 (1.74)
  Week 10; n = 175, 171 | 3.31 (1.53) | 3.34 (1.74)
  Week 11; n = 173, 167 | 3.23 (1.56) | 3.30 (1.77)
  Week 12; n = 172, 169 | 3.18 (1.54) | 3.21 (1.77)

4. Secondary Outcome: The Area Under the HCV-RNA Curve Estimated From the Two Adjacent Pre-dose Assessments at Each Week
Description: The area under the HCV-RNA curve (HCV AUC) was defined as the area under the polygonal line defined by the HCV RNA values from the beginning of the time window to the end of the time window. Each of these areas was a sum of one or more trapezoids determined from the concentrations over the 7-day interval. The HCV AUC to Week 12 was the sum of the 12 weekly HCV AUCs divided by the time (12 weeks). Summary of weekly HCV AUC values estimated from the two adjacent pre-dose assessments are presented.
Time Frame: From Week -1 to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log 10 IU/mL
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 188 | 190
log 10 IU/mL
  Week -1, n = 188, 190 | 6.5 (0.40) | 6.5 (0.41)
  Week 1, n = 186, 188 | 6.1 (0.55) | 6.1 (0.56)
  Week 2, n = 185, 187 | 5.5 (0.97) | 5.4 (1.04)
  Week 3, n = 184, 184 | 5.0 (1.20) | 4.9 (1.33)
  Week 4, n = 183, 181 | 4.7 (1.36) | 4.4 (1.48)
  Week 5, n = 182, 181 | 4.3 (1.45) | 4.1 (1.57)
  Week 6, n = 180, 179 | 4.1 (1.48) | 3.9 (1.63)
  Week 7, n = 180, 177 | 3.8 (1.52) | 3.7 (1.66)
  Week 8, n = 178, 175 | 3.6 (1.54) | 3.6 (1.65)
  Week 9, n = 176, 173 | 3.5 (1.54) | 3.5 (1.68)
  Week 10, n = 176, 171 | 3.4 (1.54) | 3.4 (1.72)
  Week 11, n = 174, 170 | 3.3 (1.55) | 3.3 (1.73)
  Week 12, n = 171, 169 | 3.2 (1.55) | 3.2 (1.74)

5. Secondary Outcome: Mean Value of Area Under the HCV-RNA Curve Minus Baseline From Week 1 to Week 12
Description: The HCV AUC was calculated for each week as the area under the polygonal line defined by the HCV RNA values from the beginning of the time window to the end of the time window. Each of these areas was a sum of one or more trapezoids determined from the concentrations over the 7-day interval. The weekly AUCMB was calculated by subtracting the Week -1 HCV AUC (i.e., baseline) from the weekly HCV AUC and presented.
Time Frame: Baseline, Week 1 to Week 12
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log (IU*week/mL)
Groups:
- Peginterferon Alfa-2a + Ribavirin: Participants received Peginterferon alfa-2a at a dosage of 180 μg SC once a week plus Ribavirin 1000 or 1200 mg/day, orally (< or >/= 75 kg body weight, respectively) twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a180 μg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
- Peginterferon Alfa-2b + Ribavirin: Participants received Peginterferon alfa-2b at a dosage of 1.5 μg/kg SC once weekly plus Ribavirin1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily during the randomized treatment period for 12 weeks. Participants who completed the randomized treatment period of 12 weeks and wished to continue therapy were given Peginterferon alfa-2a 180 μg SC once weekly plus Ribavirin 1000 or 1200 mg/day orally (< or >/=75 kg body weight, respectively) twice daily for an additional 36 weeks to complete a full 48-week treatment course. After treatment completion, participants were followed-up for safety for 24 weeks.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 186 | 188
log (IU*week/mL)
  Week 1; n = 186, 188 | 0.4 (0.40) | 0.4 (0.43)
  Week 2; n = 185, 187 | 1.0 (0.90) | 1.1 (0.99)
  Week 3; n = 184, 184 | 1.4 (1.15) | 1.6 (1.30)
  Week 4; n = 183, 181 | 1.8 (1.33) | 2.0 (1.46)
  Week 5; n = 182, 181 | 2.1 (1.42) | 2.3 (1.56)
  Week 6; n = 180, 179 | 2.4 (1.47) | 2.6 (1.62)
  Week 7; n = 180, 177 | 2.6 (1.51) | 2.8 (1.66)
  Week 8; n = 178, 175 | 2.8 (1.53) | 2.9 (1.65)
  Week 9; n = 176, 173 | 3.0 (1.55) | 3.0 (1.69)
  Week 10; n = 176, 171 | 3.1 (1.55) | 3.1 (1.75)
  Week 11; n = 174, 170 | 3.2 (1.56) | 3.2 (1.76)
  Week 12; n = 171, 169 | 3.2 (1.56) | 3.2 (1.77)

6. Secondary Outcome: Cumulative Viral Absolute Area Under the HCV RNA Curve Minus Baseline Averaged Over the 12-week Period
Description: The area under the HCV-RNA curve (HCV AUC) was calculated for each week as the area under the polygonal line defined by the HCV RNA values from the beginning of the window to the end of the window. Each of these areas was a sum of one or more trapezoids determined from the concentrations over the 7-day interval. The weekly AUCMB was calculated by subtracting the Week -1 HCV AUC (i.e., baseline) from the weekly HCV AUC. The HCV AUCMB to Week 12 was the sum of the 12 weekly HCV AUCMBs divided by the time (12 weeks).
Time Frame: Up to Week 12
Population: The analysis population was ITT Population. The ITT Population included all participants who were randomized and received at least one dose of study medication (PEG-IFN or ribavirin).
Measure: Mean (Standard Deviation); unit: log10 IU/mL
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 171 | 169
log10 IU/mL | 26.9 (15.34) | 28.7 (16.66)
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; The treatment groups were compared using an analysis of variance (ANOVA) with treatment as the only factor in the model; Test type: Superiority or Other; p = 0.304, ANOVA

7. Secondary Outcome: Weekly Viral Absolute Area Under the HCV RNA Curve Estimated in the Frequent-sampling Cohort for Weeks 1 and 8
Description: The area under the HCV-RNA curve (HCV AUC) was defined as the area under the polygonal line defined by the HCV RNA values from the beginning of the window to the end of the window. For the frequent-sampling cohort, HCV AUCs over 7 days were calculated for Weeks 1 and 8, with intervals calculated beginning at the dose after which the frequent sampling began (different from the 7-day calendar period used for other AUC calculations). The AUCs for Weeks 1 and 8 in the frequent-sampling cohort (Sparse samples [SS] and frequent samples [FS]) were calculated using the trapezoidal rule.
Time Frame: Week 1 and Week 8
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log (IU*week/mL)
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 12 | 13
log (IU*week/mL)
  SS, Week 1; n = 12, 13 | 6.0 (0.45) | 6.0 (0.44)
  SS, Week 8; n = 12, 12 | 3.4 (1.65) | 3.5 (1.68)
  FS, Week 1; n = 12, 13 | 5.8 (0.52) | 5.5 (0.91)
  FS, Week 8; n = 12, 12 | 3.3 (1.63) | 3.5 (1.60)

8. Secondary Outcome: Percentage of Participants With a ≥ 2-log10 Decrease or Undetectable (< 60 International Units Per Milliliter) HCV RNA at Each Visit
Description: The virological response was determined as the proportion/percentage of participants with a ≥ 2-log10 decrease or undetectable HCV RNA at each week. Detection of >= 2-log10 decrease of <60 IU/mL HCV-RNA was done by amplicor PCR assay at each week. Detection of >=2-log10 decrease or undetectable HCV RNA at Week 12 was considered an early virological response (EVR).
Time Frame: From Week 1 to Week 12
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 189 | 191
percentage of participants
  Week 1 | 6.9 [3.3 to 10.5] | 9.9 [5.7 to 14.2]
  Week 2 | 20.1 [14.4 to 25.8] | 30.4 [23.8 to 36.9]
  Week 3 | 31.7 [25.1 to 38.4] | 42.4 [35.4 to 49.4]
  Week 4 | 41.8 [34.8 to 48.8] | 49.2 [42.1 to 56.3]
  Week 5 | 46.6 [39.4 to 53.7] | 53.4 [46.3 to 60.5]
  Week 6 | 53.4 [46.3 to 60.6] | 55.5 [48.4 to 62.5]
  Week 7 | 57.1 [50.1 to 64.2] | 57.6 [50.6 to 64.6]
  Week 8 | 61.4 [54.4 to 68.3] | 59.2 [52.2 to 66.1]
  Week 9 | 59.8 [52.8 to 66.8] | 57.6 [50.6 to 64.6]
  Week 10 | 65.6 [58.8 to 72.4] | 60.2 [53.3 to 67.2]
  Week 11 | 65.1 [58.3 to 71.9] | 59.7 [52.7 to 66.6]
  Week 12 | 66.1 [59.4 to 72.9] | 63.4 [56.5 to 70.2]
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 1: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.2814, Chi-squared; Difference in proportion of participants = -3.1, 95% CI 2-sided [-8.6 to 2.5]
Statistical Analysis 2: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 2: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.0214, Chi-squared; Difference in proportion of participants = -10.3, 95% CI 2-sided [-18.9 to -1.6]
Statistical Analysis 3: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 3: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.0315, Chi-squared; Difference in proportion of participants = -10.7, 95% CI 2-sided [-20.3 to -1.0]
Statistical Analysis 4: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 4: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.1467, Chi-squared; Difference in proportion of participants = -7.4, 95% CI 2-sided [-17.4 to 2.6]
Statistical Analysis 5: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 5: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.1823, Chi-squared; Difference in proportion of participants = -6.8, 95% CI 2-sided [-16.9 to 3.2]
Statistical Analysis 6: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 6: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.6871, Chi-squared; Difference in proportion of participants = -2.1, 95% CI 2-sided [-12.1 to 8.0]
Statistical Analysis 7: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 7: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.9295, Chi-squared; Difference in proportion of participants = -0.4, 95% CI 2-sided [-10.4 to 9.5]
Statistical Analysis 8: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 8: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.6593, Chi-squared; Difference in proportion of participants = 2.2, 95% CI 2-sided [-7.6 to 12.1]
Statistical Analysis 9: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 9: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.6637, Chi-squared; Difference in proportion of participants = 2.2, 95% CI 2-sided [-7.7 to 12.1]
Statistical Analysis 10: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 10: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.2760, Chi-squared; Difference in proportion of participants = 5.4, 95% CI 2-sided [-4.3 to 15.1]
Statistical Analysis 11: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 11: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.2779, Chi-squared; Difference in proportion of participants = 5.4, 95% CI 2-sided [-4.3 to 15.1]
Statistical Analysis 12: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 12: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.5697, Chi-squared; Difference in proportion of participants = 2.8, 95% CI 2-sided [-6.8 to 12.4]

9. Secondary Outcome: Percentage of Participants With Undetectable HCV RNA (< 60 International Units/Milliliter) at Each Visit
Description: The viral load was determined quantitatively and qualitatively by HCV-polymerase chain reaction (PCR). Qualitative viral titers will be assessed by Roche amplicor HCV Monitor® test v2.0 (< 600 IU/mL). The virological response was determined as the percentage of participants with undetectable HCV RNA at each week. A <60 IU/mL HCV-RNA was measured by amplicor PCR assay.
Time Frame: From Week 1 to Week 12
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 189 | 191
percentage of participants
  Week 1 | 0.5 [-0.5 to 1.6] | 0.5 [-0.5 to 1.5]
  Week 2 | 1.6 [-0.2 to 3.4] | 2.1 [0.1 to 4.1]
  Week 3 | 2.6 [0.4 to 4.9] | 6.3 [2.8 to 9.7]
  Week 4 | 7.4 [3.7 to 11.1] | 11.5 [7.0 to 16.0]
  Week 5 | 11.1 [6.6 to 15.6] | 15.7 [10.5 to 20.9]
  Week 6 | 16.9 [11.6 to 22.3] | 23.6 [17.5 to 29.6]
  Week 7 | 22.2 [16.3 to 28.1] | 26.7 [20.4 to 33.0]
  Week 8 | 25.9 [19.7 to 32.2] | 29.3 [22.9 to 35.8]
  Week 9 | 29.6 [23.1 to 36.1] | 35.6 [28.8 to 42.4]
  Week 10 | 34.9 [28.1 to 41.7] | 40.3 [33.4 to 47.3]
  Week 11 | 39.2 [32.2 to 46.1] | 41.9 [34.9 to 48.9]
  Week 12 | 39.2 [32.2 to 46.1] | 44.0 [36.9 to 51.0]
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 1: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.9940, Chi-squared; Difference in proportion of participants = 0.0, 95% CI 2-sided [-1.4 to 1.5]
Statistical Analysis 2: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 2: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.7133, Chi-squared; Difference in proportion of participants = -0.5, 95% CI 2-sided [-3.2 to 2.2]
Statistical Analysis 3: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 3: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.0864, Chi-squared; Difference in proportion of participants = -3.6, 95% CI 2-sided [-7.8 to 0.5]
Statistical Analysis 4: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 4: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.1713, Chi-squared; Difference in proportion of participants = -4.1, 95% CI 2-sided [-10.0 to 1.8]
Statistical Analysis 5: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 5: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.1888, Chi-squared; Difference in proportion of participants = -4.6, 95% CI 2-sided [-11.4 to 2.2]
Statistical Analysis 6: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 6: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.1080, Chi-squared; Difference in proportion of participants = -6.6, 95% CI 2-sided [-14.7 to 1.4]
Statistical Analysis 7: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 7: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.3099, Chi-squared; Difference in proportion of participants = -4.5, 95% CI 2-sided [-13.1 to 4.2]
Statistical Analysis 8: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 8: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.4595, Chi-squared; Difference in proportion of participants = -3.4, 95% CI 2-sided [-12.4 to 5.6]
Statistical Analysis 9: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 9: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.2144, Chi-squared; Difference in proportion of participants = -6.0, 95% CI 2-sided [-15.4 to 3.4]
Statistical Analysis 10: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 10: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.2779, Chi-squared; Difference in proportion of participants = -5.4, 95% CI 2-sided [-15.1 to 4.3]
Statistical Analysis 11: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 11: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.5876, Chi-squared; Difference in proportion of participants = -2.7, 95% CI 2-sided [-12.6 to 7.1]
Statistical Analysis 12: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 12: Treatment groups were compared using the Chi-Square Test; Test type: Superiority or Other; p = 0.3399, Chi-squared; Difference in proportion of participants = -4.8, 95% CI 2-sided [-14.7 to 5.1]

10. Secondary Outcome: Number of Participants With Marked Hematologic Abnormalities
Description: The values outside the marked reference range for any hematology parameter that represents a defined, clinically relevant change from baseline are considered marked hematology abnormalities. The Roche standard reference ranges for the hematology parameters for which subjects had marked abnormalities were hematocrit [(RR) is 0.42 - 0.52 (fraction)], hemoglobin (RR is 13.0 - 18.0 gram/deciliter), platelets (RR is 150 - 450 10^9 cells/L), white blood cells (WBC) (RR is 4.3 - 10.8 10^9 cells/L), basophils (RR is 0.00 - 0.15 10^9 cells/L), lymphocytes (RR is 1.50 - 4.00 10^9 cells/L), monocytes (RR is 0.20 - 0.95 10^9 cells/L), neutrophils (RR is 1.83 - 7.25 10^9 cells/L), prothrombin time (PT) (RR is 9 - 13 seconds), partial thromboplastin time (Partial Throm.) (Time) (RR is 25.0 - 38.0 seconds) and PT International normalized ratio (INR) [RR is 0.70 - 1.30 (ratio)]. Summary data of number of participants with only marked hematology abnormalities are presented.
Time Frame: Baseline, up to Week 12
Population: The analysis population was the Safety Population. The Safety Population included all participants who were randomized, received at least one dose of study medication (PEG-IFN or ribavirin), and had at least one post-baseline safety assessment (defined as clinical adverse event, laboratory or vital sign data, or physical examination finding).
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 187 | 190
participants
  Hemoglobin-Low | 64 | 69
  Platelets-Low | 41 | 31
  Hematocrit -Low | 72 | 90
  WBC-High | 2 | 0
  WBC-Low | 124 | 119
  Basophils-High | 2 | 0
  Lymphocytes-Low | 77 | 75
  Monocytes-Low | 1 | 1
  Neutrophils-Low | 136 | 137
  Partial Throm.-High | 3 | 1
  PT (ProThrom Time)-High | 15 | 25
  PT (INR)-High | 5 | 6

11. Secondary Outcome: Number of Participants With Marked Biochemical Test Abnormalities
Description: Values outside the marked RR for biochemical test parameters that represent a defined, clinically relevant change from baseline are considered marked biochemical test abnormalities. Roche's standard RR for biochemical parameters were used for this analysis. The biochemical test parameters with marked abnormalities were alanine aminotransferase (ALAT) (RR is 0 - 30 units per liter [U/L]), aspartate aminotransferase (ASAT) (RR is 0 - 25 U/L), gamma-glutamyl transferase (GGT) (RR is 0 - 60 U/L), total bilirubin (RR is 0 - 17 micromole/liter [umol/L]), creatinine (RR is 0 - 133 umol/L), total protein (RR is 60 - 80 g/L), triglycerides (RR is 0.45 - 1.70 millimole/liter [mmol/L]), chloride (RR is 100 - 108 mmol/L), potassium (RR is 3.5 - 5.0 mmol/L), sodium (RR is 133 - 145 mmol/L), calcium (RR is 2.10 - 2.60 mmol/L), random glucose (RR is 3.89 - 7.83 mmol/L), uric acid (140 - 500 umol/L). Summary data of number of participants with only marked biochemical test abnormalities are presented.
Time Frame: Baseline, up to Week 12
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 187 | 190
participants
  ALAT-High | 5 | 12
  ASAT- High | 17 | 11
  GG- High | 23 | 18
  Total Bilirubin- High | 8 | 8
  Creatinine- High | 0 | 1
  Total Protein- Low | 1 | 4
  Triglycerides- High | 89 | 98
  Chloride- Low | 2 | 5
  Potassium- Low | 1 | 2
  Sodium- Low | 1 | 5
  Calcium- Low | 5 | 9
  Glucose Random- High | 3 | 5
  Uric Acid- High | 8 | 21

12. Secondary Outcome: Number of Participants With Marked Abnormalities in Thyroid Function Tests
Description: Values outside the marked reference ranges for thyroid function test parameters that represent a defined, clinically relevant change from baseline are considered marked thyroid function test abnormalities. Roche's standard reference ranges for thyroid function test parameters were used for the analysis. The thyroid function parameters with marked abnormalities were triiodothyronine (T3) (RR is 1.20 - 3.00 nanomole/liter [nmol/L]), thyroxine (T4) (RR is 51 - 154 nmol/L) and thyroid stimulating hormone (TSH) (RR is 0.0 - 5.0 milliunits per liter [mU/L]). Summary data of number of participants with only marked abnormalities in thyroid function tests are presented.
Time Frame: Baseline, up to Week 12
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 187 | 190
participants
  T3-High | 4 | 3
  T4-High | 4 | 2
  TSH-High | 1 | 1

13. Secondary Outcome: Mean Trough Interferon Concentrations at Each Week
Description: The weekly Interferon (IFN) concentrations were calculated using the trapezoid rule. The trough IFN concentration was analyzed using an enzyme-linked immunosorbent assay (ELISA), with limits of quantification of 250 picograms per milliliter [pg/mL] for Pegasys and 150 pg/mL for PEG-Intron respectively.
Time Frame: From Week 1 to Week 12
Population: as for outcome 3
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 152 | 182
pg/mL
  Week 1; n = 137, 179 | 6730 (289.3) | 119 (11.0)
  Week 2; n = 152, 182 | 9530 (399.6) | 144 (12.1)
  Week 3; n = 152, 181 | 11082 (438.4) | 125 (8.8)
  Week 4; n = 152, 178 | 12089 (439.0) | 150 (16.7)
  Week 5; n = 150, 177 | 12529 (454.7) | 163 (16.2)
  Week 6; n = 150, 173 | 12686 (429.9) | 143 (10.4)
  Week 7; n = 150, 175 | 12852 (438.8) | 162 (14.6)
  Week 8; n = 146, 174 | 12781 (448.3) | 147 (10.4)
  Week 9; n = 144, 171 | 12781 (422.2) | 167 (17.3)
  Week 10; n = 145, 168 | 12499 (397.3) | 156 (12.2)
  Week 11; n = 144, 165 | 12689 (409.2) | 163 (10.9)
  Week 12; n = 144, 168 | 12846 (450.9) | 154 (11.4)

14. Secondary Outcome: Area Under the Curve for Interferon in the Frequent-Sampling Cohort
Description: Area Under the Curve (AUC) for Interferon (IFN) for Week 1 and Week 8 in the frequent-sampling cohort were calculated using the trapezoidal rule.
Time Frame: Week 1 and Week 8
Population: The analysis population was ITT Population. The ITT Population included all participants who were randomized and received at least one dose of study medication (PEG-IFN or ribavirin). The "n" represents the number of participants assessed for AUC for Interferon for specified time point.
Measure: Mean (Standard Deviation); unit: week*pg/mL
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 8 | 5
week*pg/mL
  Week 1; n = 8, 4 | 6376.0 (2551.53) | 315.2 (79.39)
  Week 8; n = 7, 5 | 14399.9 (5658.05) | 472.1 (62.32)
Statistical Analysis 1: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 1: The treatment groups were compared using repeated measures analysis; Test type: Superiority or Other; p = 0.024, Repeated measures analysis; The P-value is determined from a repeated measures analysis with terms for treatment group, baseline, week, and the week-by-treatment interaction
Statistical Analysis 2: Comparison: Peginterferon Alfa-2a + Ribavirin vs Peginterferon Alfa-2b + Ribavirin; Week 8: The treatment groups were compared using Repeated measures analysis; Test type: Superiority or Other; p < 0.001, Repeated measures analysis

15. Secondary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject who is administered a study treatment regardless of whether or not the event has a causal relationship with the treatment. An AE, therefore, could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the study treatment, whether or not related to the treatment. A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect. Number of participants with at least one AE and SAE were reported.
Time Frame: Up to Week 12
Population: as for outcome 10
Measure: Number; unit: participants
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 187 | 190
participants
  Any AE | 185 | 187
  Any SAE | 5 | 2

16. Secondary Outcome: Percentage of Participants With Each of the Identified HCV Quasispecies at Baseline and Weeks 1, 4, 8, and 12
Description: The determination of evolution of HCV quasispecies in participants was planned through analyzing viral sequences in serum samples drawn at baseline and at Weeks 1, 4, 8, and 12 if HCV RNA tests were positive and if the levels were sufficient to do the analysis.
Time Frame: Baseline, Weeks 1, 4,8, and 12
Population: The ITT Population included all participants who were randomized and received at least one dose of study medication (PEG-IFN or ribavirin). This outcome measure was not analyzed as no data were collected for any of the participants in this study.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Weekly AUC for IFN Concentrations for Pegasys and PEG-Intron Estimated by Population Pharmacokinetic Modeling
Description: The estimation of weekly AUC for IFN concentrations for Pegasys and PEG-Intron was planned through population pharmacokinetic modeling. A population pharmacokinetic method deals with modelling in a cohort which has many participants (usually more than 40). The estimation of weekly AUC for IFN concentrations for Pegasys and PEG-Intron was planned to be studied in the population rather than the individuals in Peginterferon alfa-2a + Ribavirin and Peginterferon alfa-2b + Ribavirin groups.
Time Frame: Up to Week 8
Population: as for outcome 16
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 72
Description: The adverse events were reported in safety population (187 and 190 participants in Peginterferon Alfa-2a + Ribavirin and Peginterferon Alfa-2b + Ribavirin respectively). The non-serious AEs were reported only till Week 12.
Arm/Group | Peginterferon Alfa-2a + Ribavirin | Peginterferon Alfa-2b + Ribavirin
Serious Adverse Events (participants affected / at risk) | 14/187 | 16/190
Other Adverse Events (participants affected / at risk) | 184/187 | 186/190
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=187) | Peginterferon Alfa-2b + Ribavirin (N=190)
Colitis ischaemic (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 2 | 1
Pelvic mass (General disorders) | 1 | 1
Pneumonia (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Viral rash (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Syncope (Nervous system disorders) | 0 | 3
Hemiparesis (Nervous system disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1
Mania (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginterferon Alfa-2a + Ribavirin (N=187) | Peginterferon Alfa-2b + Ribavirin (N=190)
Fatigue (General disorders) | 133 | 137
Chills (General disorders) | 46 | 79
Irritability (General disorders) | 58 | 57
Pyrexia (General disorders) | 38 | 62
Influenza like illness (General disorders) | 34 | 44
Injection site erythema (General disorders) | 25 | 38
Pain (General disorders) | 25 | 28
Injection site rash (General disorders) | 8 | 17
Nausea (Gastrointestinal disorders) | 77 | 85
Diarrhoea (Gastrointestinal disorders) | 39 | 40
Vomiting (Gastrointestinal disorders) | 26 | 38
Dyspepsia (Gastrointestinal disorders) | 14 | 18
Abdominal pain (Gastrointestinal disorders) | 16 | 12
Constipation (Gastrointestinal disorders) | 11 | 17
Dry mouth (Gastrointestinal disorders) | 9 | 18
Abdominal pain upper (Gastrointestinal disorders) | 8 | 13
Headache (Nervous system disorders) | 105 | 113
Dizziness (Nervous system disorders) | 39 | 48
Dysguesia (Nervous system disorders) | 17 | 21
Disturbance in attention (Nervous system disorders) | 11 | 17
Insomnia (Psychiatric disorders) | 69 | 69
Depression (Psychiatric disorders) | 46 | 49
Anxiety (Psychiatric disorders) | 18 | 17
Rash (Skin and subcutaneous tissue disorders) | 27 | 42
Pruritis (Skin and subcutaneous tissue disorders) | 28 | 30
Dry skin (Skin and subcutaneous tissue disorders) | 25 | 31
Alopecia (Skin and subcutaneous tissue disorders) | 6 | 13
Rash pruritic (Skin and subcutaneous tissue disorders) | 10 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 44 | 41
Myalgia (Musculoskeletal and connective tissue disorders) | 31 | 34
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 17 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 29 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 | 23
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 14 | 17
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 11
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 13
Decreased appetite (Metabolism and nutrition disorders) | 28 | 40
Anorexia (Metabolism and nutrition disorders) | 18 | 24
Vision blurred (Eye disorders) | 8 | 18
Dry eye (Eye disorders) | 6 | 12
Anaemia (Blood and lymphatic system disorders) | 20 | 22
Upper respiratory tract infection (Infections and infestations) | 10 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights